CLINICAL TRIAL: NCT02683109
Title: A 4-week, Randomised, Double-blind, Parallel Group Study to Evaluate the Efficacy and Safety of Tiotropium + Olodaterol Fixed Dose Combination (5/5 µg) Delivered by the Respimat® Inhaler Versus the Free Combination of Tiotropium 5 µg and Olodaterol 5 µg Delivered by Separate Respimat® Inhalers in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Fixed Dose Combination Versus Free Combination of Tiotropium and Olodaterol in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.49; 2015-003879-29 (EudraCT Number)
Record Dates: First submitted 2016-02-12; First posted 2016-02-17 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- FDC of tiotropium + olodaterol (Experimental): Fixed Dose Combination of tiotropium + olodaterol
  Interventions: Drug: FDC of tiotropium + olodaterol; Drug: Placebo
- Free combination tiotropium + olodaterol (Active Comparator)
  Interventions: Drug: Tiotropium; Drug: Olodaterol

INTERVENTIONS:
Drug: FDC of tiotropium + olodaterol — Fixed Dose Combination of tiotropium + olodaterol
  Arms: FDC of tiotropium + olodaterol
Drug: Placebo
  Arms: FDC of tiotropium + olodaterol
Drug: Tiotropium
  Arms: Free combination tiotropium + olodaterol
Drug: Olodaterol
  Arms: Free combination tiotropium + olodaterol

SUMMARY:
This is a 4-week, multicenter, randomized, double-blind, parallel group and active controlled study.

Patients will be randomized (1 to 1 ratio) to a 4-week double-blind treatment period of either FDC (fixed-dose combination) of tiotropium + olodaterol (5/5 µg) plus placebo or the free combination of tiotropium 5 µg and olodaterol 5 µg; all administered via the Respimat® inhaler. The purpose is to show non-inferiority between the FDC and the free combination of tiotropium and olodaterol in patients with COPD.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients.
* Patients 40 years of age or older.
* Patients with a smoking history > 10 pack years.
* Diagnostic of COPD with Post-bronchodilator FEV1 (Forced Expiratory Volume in one second) >= 30% and <80% of predicted normal and Post-bronchodilator FEV1/FVC (Forced Vital Capacity) <70% at screening.
* Symptomatic patients with CAT (COPD Assessment Test TM) score >= 10 at screening.
* Further inclusion criteria apply.

Exclusion criteria:

* COPD exacerbation or symptoms of lower respiratory tract infection within 6 weeks prior to screening.
* Patients with a current diagnosis of asthma.
* Further exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (22):
- Austria (2):
  - Ordination Dr. Robert Voves, 8330 Feldbach, Feldbach
  - KH d. Elisabethinen Linz, Linz
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus
  - Hvidovre Hospital, Hvidovre
  - Regionshospitalet Silkeborg, Silkeborg
- Finland (5):
  - Jorvin sairaala, Espoo
  - HYKS Keuhkosairauksien, Helsinki
  - TAYS, Keuhkotautien poliklinikka, Tampere
  - TYKS, Keuhkosairauksien klinikka, Turku, Turku
  - Terveystalo Pulssi, Turku, Turku
- France (9):
  - HOP Louis Pradel, Bron
  - CLI du Parc, Pneumo, Castelnau le Lez, Castelnau-le-Lez
  - CAB Pigearias B., Pneumo, Nice, Nice
  - CAB Dupouy J, Pneumo, Nîmes, Nîmes
  - HOP Cochin, Paris
  - HOP Haut-Lévêque, Pessac
  - HOP Maison Blanche, Reims
  - INS A.Tzanck,Pneumo,St Laurent du Var, Saint-Laurent-du-Var
  - CAB Lejay D, MG, Vieux Condé, Vieux-Condé
- Slovenia (3):
  - Univ. Clinic of Respiratory and Allergic Diseases, Golnik, Golnik
  - Verboten Kopriva Renata - Private practice, Litija, Litija
  - Arjana Macek d.o.o., Ljubljana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Definition: Open-Label Treated Set (OLTS): This patient set includes all patients who signed the informed consent and were dispensed open-label study medication during the run-in period prior to randomisation and were documented to have taken any dose of this medication.
Pre-assignment Details: Definition: Randomised Set (RS): This patient set is nested within the OLTS and includes all patients who signed the informed consent form and were also randomised, regardless of whether the patient was treated with study medication or not.
Groups:
- T+O 5/5: The subjects were administered Tiotropium (T) + Olodaterol (O) Fixed Dose Combination (FDC) solution for inhalation 2.5 μg/2.5 μg per actuation, 2 inhalations orally once daily via RESPIMAT® inhaler.
  Placebo matching Tiotropium solution was administered 2 inhalations once daily via RESPIMAT® inhaler.
- T 5/O 5: The subjects were administered Tiotropium solution for inhalation, 2.5 μg per actuation + Olodaterol solution for inhalation, 2.5 μg per actuation as a free combination. Two inhalations were administered once daily (a.m. dosing) via RESPIMAT® inhaler for both Tiotropium and Olodaterol.
Period: Overall Study
Arm/Group | T+O 5/5 | T 5/O 5
Started | 110 | 111
Completed | 109 | 111
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set [TS]: This patient set is nested within the RS and includes all patients who were dispensed study medication and were documented to have taken any dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | T+O 5/5 | T 5/O 5 | Total
Number analyzed (Participants) | 110 | 111 | 221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (7.1) | 66.5 (6.4) | 66.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 63
  Male | 77 | 81 | 158

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) (in Liter) After 28 Days of Treatment
Description: This outcome measure presents FEV1 after 28 days of treatment (measurement on Day 29). Trough FEV1 was defined as the FEV1 value at the end of the dosing interval (24 hours), and was measured at 24 hours (+/- 10 minutes) after trial medication administration at Visit 5.
  The FEV1 measurement at Visit 4, which was 24 hours after the last open-label run-in treatment intake and 15 minutes before the first double-blind study drug intake was the baseline measurement.
Time Frame: Day 29
Population: Full Analysis Set (FAS): This patient set is nested within the TS and includes patients who had a baseline measurement and at least one post-baseline measurement for the primary endpoint.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | T+O 5/5 | T 5/O 5
Number analyzed (Participants) | 108 | 108
Liter | 1.422 (0.016) | 1.399 (0.016)
Statistical Analysis 1: Comparison: T+O 5/5 vs T 5/O 5; The primary analysis was conducted using an Analysis of Covariance [ANCOVA] model including treatment as fixed categorical effect and baseline as continuous covariate; Test type: Non-Inferiority or Equivalence — Non-inferiority of the Tio+Olo FDC versus the Tio/Olo free combination was tested at the one-sided α-level of 0.025 using a non-inferiority margin of 0.1 L; p < 0.0001, ANCOVA; Adjusted mean = 0.024, 95% CI 2-sided [-0.020 to 0.067], Standard Error of Mean 0.022

2. Secondary Outcome: Trough Forced Vital Capacity (FVC) (in Liter) After 28 Days of Treatment
Description: This outcome measure presents trough FVC after 28 days of treatment (measurement on Day 29).
  The FVC measurement at Visit 4, which was 24 hours after the last open-label run-in treatment intake and 15 minutes before the first double-blind study drug intake was the baseline measurement for FVC.
Time Frame: Day 29
Population: FAS.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | T+O 5/5 | T 5/O 5
Number analyzed (Participants) | 108 | 108
Liter | 3.126 (0.024) | 3.121 (0.024)
Statistical Analysis 1: Comparison: T+O 5/5 vs T 5/O 5; The secondary analysis was conducted using an ANCOVA model including treatment as fixed categorical effect and baseline as continuous covariate; Test type: Superiority or Other; p = 0.8648, ANCOVA; Adjusted mean = 0.006, 95% CI 2-sided [-0.061 to 0.073], Standard Error of Mean 0.034

3. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Assessment Test™ (CAT) Score on Day 28
Description: This outcome measure presents COPD assessment test score on Day 28. The COPD Assessment Test™ is a short 8-item questionnaire for assessment and monitoring of COPD health status in routine practice. Its scale is 0-40 (high score = poor health).
  The CAT measurement on Visit 4 prior to the first dose of double-blind study drug was the baseline for CAT.
Time Frame: Day 28
Population: FAS. One patient in the T 5/O 5 free combination group had missing data for the CAT questionnaire.
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | T+O 5/5 | T 5/O 5
Number analyzed (Participants) | 108 | 107
Score on scale | 15.423 (0.377) | 15.750 (0.379)
Statistical Analysis 1: Comparison: T+O 5/5 vs T 5/O 5; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5420, ANCOVA; Adjusted mean = -0.327, 95% CI 2-sided [-1.384 to 0.729], Standard Error of Mean 0.536

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after last drug administration, up to 49 days.
Groups:
- Total: The total number of subjects who were administered T+O 5/5 or T 5/O 5.
Arm/Group | T+O 5/5 | T 5/O 5 | Total
Serious Adverse Events (participants affected / at risk) | 1/110 | 2/111 | 3/221
Other Adverse Events (participants affected / at risk) | 9/110 | 9/111 | 18/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T+O 5/5 (N=110) | T 5/O 5 (N=111) | Total (N=221)
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T+O 5/5 (N=110) | T 5/O 5 (N=111) | Total (N=221)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.